CLINICAL TRIAL: NCT07040787
Title: A Single-center, Single-arm, Fixed-sequence Drug-drug Interaction Study of HRS-5965 With Clopidogrel and Clarithromycin in Healthy Subjects
Brief Title: Investigation of Drug-drug Interaction of HRS-5965 With Clopidogrel and Clarithromycin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chengdu Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRS-5965-107
Record Dates: First submitted 2025-06-18; First posted 2025-06-27 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Complement Mediated Glomerular Diseases; Hemolytic Anemia
MeSH Terms: conditions — Anemia, Hemolytic | interventions — Clopidogrel; Clarithromycin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug-drug interaction between HRS-5965 and clopidogrel (Experimental)
  Interventions: Drug: HRS-5965 Capsules; Drug: Clopidogrel
- Drug-drug interaction between HRS-5965 and clarithromycin (Experimental)
  Interventions: Drug: HRS-5965 Capsules; Drug: Clarithromycin

INTERVENTIONS:
Drug: HRS-5965 Capsules — Oral HRS-5965 capsules.
Drug: Clopidogrel — Oral clopidogrel.
  Arms: Drug-drug interaction between HRS-5965 and clopidogrel
Drug: Clarithromycin — Oral clarithromycin.
  Arms: Drug-drug interaction between HRS-5965 and clarithromycin

SUMMARY:
The study is being conducted to compare the drug-drug interaction of HRS-5965 with clopidogrel and clarithromycin in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the study procedures and methods, participate voluntarily and be able to complete the study according to the protocol requirements, and sign the informed consent form (ICF) in writing.
2. Aged 18-45 years old on the date of signing the ICF (including the threshold), both male and female.
3. At the time of screening, male subjects weighing no less than 50 kg and female subjects weighing no less than 45 kg; body mass index (BMI): 19~26 kg/m2 (including the threshold).
4. During the screening period, human immunodeficiency virus antibody (HIV-Ab), treponema pallidum antibody, hepatitis B surface antigen (HBsAg) and hepatitis C virus antibody (HCV-Ab) were all negative.
5. Female subjects with reproductive capacity or male subjects whose partners are female subjects with reproductive capacity need to have no plans for fertility or sperm/egg donation within 3 months +1 week for male subjects and 6 months +1 week for female subjects from the date of signing the informed consent form until the last medication use, and voluntarily take efficient contraceptive measures (including partners).

Exclusion Criteria:

1. Allergic to two or more allergens, or in the judgment of the investigator, may be allergic to the study drug or its components.
2. Disease or medical condition that, in the judgment of the investigator, may interfere with the absorption, distribution, metabolism, and excretion of the drug or that may reduce compliance.
3. Patients with a previous history of coronary artery disease, severe cardiac insufficiency, conduction disorders or clinically significant bradycardia.
4. Patients with a history of electrolyte disorders (such as hypomagnesemia).
5. Patients with a history of congenital or acquired QT interval prolongation or ventricular arrhythmia.
6. Those with a history of meningococcal infection and streptococcus pneumoniae infection.
7. Those with a history of neuromuscular diseases (such as myotonic dystrophy, poliomyelitis, myasthenia gravis, botulism poisoning) and poliomyelitis.
8. Subjects who have had or are currently suffering from active pathological bleeding.
9. Subjects with a previous history of recurrent oral ulcers.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-07-08 (Actual); Primary Completion 2025-08-17 (Actual); Study Completion 2025-08-17 (Actual)

PRIMARY OUTCOMES:
The maximum plasma concentration (Cmax) | Day 1 to day 12.
Area under the concentration curve from time 0 to the last quantifiable concentration (AUClast) | Day 1 to day 12.

SECONDARY OUTCOMES:
Time to maximum plasma concentration | Day 1 to day 12.
Terminal half-life (t1/2) | Day 1 to day 12.
Incidence and severity of adverse events (AEs) | Day 1 up to day 19.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided